CLINICAL TRIAL: NCT00900432
Title: Immune Studies of Peripheral Blood From Patients With Malignant Disease Gastrointestinal Tract
Brief Title: Immune Response in Peripheral Blood of Patients With Colon Cancer
Status: Completed | Type: Observational
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 04-0331-01; P50CA095060 (NIH); P30CA023074 (NIH); UARIZ-04-81 (Other: CDR0000491215)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2012-08

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Immunoenzyme Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: immunoenzyme technique
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that may occur in the immune system that may help kill cancer cells.

PURPOSE: This laboratory study is looking at anticancer immune responses in the peripheral blood of patients with colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Quantify T cells specific for tumor peptides (carcinoembryonic antigen and MUC1) from the peripheral blood of patients with colon cancer.

OUTLINE: This is an open-label study.

Patients undergo blood collection at time of follow-up, surgery, thoracentesis, paracentesis, or leukapheresis (≤ 5 times per year). Blood is analyzed for tumor peptides (carcinoembryonic antigen and MUC1), circulating cytokines, and lymphocyte response by ELISA, ELISPOT, or intracellular flow.

PROJECTED ACCRUAL: A total of 140 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of colon cancer

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: colon cancer
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2004-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Quantitation of T cells specific for tumor peptides (carcinoembryonic antigen and MUC1) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Demeure, MD, Study Chair — University of Arizona
Locations (1):
- Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona, United States